CLINICAL TRIAL: NCT05275855
Title: A First-in-human, Randomized, Participant and Investigator Blinded, Placebo Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of EDI048 in Healthy Volunteers
Brief Title: First in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of EDI048 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CEDI048A02101
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: EDI048 or Placebo (Experimental): Part A is a single ascending dose study
  Interventions: Drug: EDI048; Other: Placebo
- Part B: EDI048 or Placebo (Experimental): Part B is a multiple ascending dose study
  Interventions: Drug: EDI048; Other: Placebo

INTERVENTIONS:
Drug: EDI048 — Oral Liquid
Other: Placebo — Oral Liquid

SUMMARY:
A first-in-human study to evaluate the safety, tolerability, and pharmacokinetics of single ascending doses and multiple ascending doses of EDI048 administered orally in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants 18 to 55 years of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Participants must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18.0 - 30.0 kg/m2. BMI = Body weight (kg) / [Height (m)]2
* At screening and baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the supine position after the participant has rested for at least three (3) minutes, and again in the standing position. Supine vital signs should be within the following ranges:
* oral body temperature between 35.0-37.5 °C
* systolic blood pressure, 90-139 mmHg
* diastolic blood pressure, 50-89 mmHg
* pulse rate, 40-90 bpm

Exclusion Criteria:

* Participants who have received any IMP in a clinical research study within 90 days or 5 half-lives of enrollment, whichever is longer; or longer if required by local regulations.
* History of multiple and recurring allergies or allergy or hypersensitivity to any of the study treatments, excipients or drugs of similar chemical classes. Hay fever is allowed unless it is active at time of screening or if there is a risk that it may become active during the study.
* Pregnant or nursing (lactating) women, assessed at screening and baseline.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Sexually active males unwilling to use a condom during intercourse while taking investigational drug and for 7 days after stopping the investigational drug.

Additional protocol-defined inclusion / exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 8.5 weeks for Part A and 9 weeks for Part B
  Number of participants with AEs and Serious Adverse Events (AEs), including significant changes from baseline in vital signs, electrocardiograms and laboratory assessments qualifying and reported as AEs.

SECONDARY OUTCOMES:
Parts A and B: Cmax | up to 13 days
  Characterize the Cmax profile following EDI048 dosing
Parts A and B: Tmax | up to 13 days
  Characterize the Tmax profile following EDI048 dosing
Parts A and B: AUClast | up to 13 days
  Characterize the AUClast profile following EDI048 dosing
Parts A and B: AUCinf | up to 13 days
  Characterize the AUCinf profile following EDI048 dosing
Parts A and B: T1/2 | up to 13 days
  Characterize the T1/2 profile following EDI048 dosing
Part B: AUC0-12h | up to 13 days
  Characterize the AUC0-12h profile following EDI048 dosing
Part B: Accumulation (Racc) | up to 13 days
  Characterize the Racc profile following EDI048 dosing
Part A: Renal Clearance (CLr) | up to 13 days
  Characterize the CLr profile following EDI048 dosing
Part A: Ae0-t | up to 3 day
  Assess amount of EDI048 excreted in urine

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Mere Way, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No